CLINICAL TRIAL: NCT03327025
Title: Survivor Health and Resilience Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013-0550
Record Dates: First submitted 2017-10-24; First posted 2017-10-31 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Pediatric Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Behavioral: Health education counseling

INTERVENTIONS:
Behavioral: Health education counseling — Health education counseling

SUMMARY:
An intervention to assist pediatric cancer survivors to behaviorally manage late effects.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric cancer survivor

Exclusion Criteria:

-

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2013-07-19 (Actual); Primary Completion 2017-03-29 (Actual); Study Completion 2017-03-29 (Actual)

PRIMARY OUTCOMES:
Tobacco use | 1 Month

IPD SHARING:
Plan to Share IPD: No